CLINICAL TRIAL: NCT02662387
Title: Use of External Nasal Dilator as an Adjuvant to High-Flow Nasal Cannula Oxygen Therapy in Children With Acute Respiratory Failure: A Prospective Randomized Controlled Trial
Brief Title: External Nasal Dilator and Oxygen Therapy in Respiratory Failure
Acronym: HFNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Janeth Chiaka Ejike, MD, Associate Professor, Pediatrics, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5150128
Record Dates: First submitted 2015-09-01; First posted 2016-01-25 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Acute Respiratory Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High flow nasal cannula (HFNC) (Active Comparator): Non-invasive positive pressure ventilation
  Interventions: Other: High flow nasal cannula (HFNC)
- HFNC and external nasal dilator (END) (Experimental): high flow nasal cannula and external nasal dilator
  Interventions: Device: External nasal dilator (END); Other: High flow nasal cannula (HFNC)

INTERVENTIONS:
Device: External nasal dilator (END) — Applying External nasal dilator as adjuvant to high flow oxygen
  Other Names: nasal strip
  Arms: HFNC and external nasal dilator (END)
Other: High flow nasal cannula (HFNC) — Non-invasive positive pressure ventilation

SUMMARY:
Acute respiratory failure secondary to bronchiolitis and asthma is one of the most common diagnoses in children admitted to pediatric intensive care unit.

Objectives: The primary outcome of the study is to compare the respiratory parameters between patients on HFNC and HFNC with ENDs.

Methods: This is a prospective randomized controlled trial. All children admitted to Loma Linda University Children's Hospital due to acute respiratory failure secondary to bronchiolitis and asthma are eligible for inclusion in the study. Multiple respiratory parameters will be collected as part of the study. The investigators anticipate that use of END will have a positive impact on the respiratory status of children with acute respiratory failure. Appropriate statistical analysis of the data will occur after the data has been de-identified.

DETAILED DESCRIPTION:
Acute respiratory failure secondary to bronchiolitis is one of the most common diagnoses in children admitted to pediatric intensive care unit.

Objectives: The primary outcome of the study is to compare the respiratory parameters between patients on high flow nasal cannula (HFNC) and HFNC with an external nasal dilator (END).

Methods: This is a prospective randomized controlled trial. All children admitted to Loma Linda University Children's Hospital between July 2015 and May 2017 for approximately 22 months due to acute respiratory failure secondary to bronchiolitis are eligible for inclusion in the study. Two arms will be studied, one with HFNC and the other with HFNC and ENDS. Modified Bronchiolitis Severity Score will be used to assess respiratory parameters as part of the study. The investigators anticipate that use of END will have a positive impact on the respiratory status of children with acute respiratory failure. Appropriate statistical analysis of the data will occur after the data has been de-identified.

ELIGIBILITY:
Inclusion Criteria:

* children less than 18years
* acute respiratory failure

Exclusion Criteria:

* immediate intubation
* >18years

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janeth Ejike, MD, Study Director — Loma Linda University Medical Center
Locations (1):
- LLUCH, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- High Flow Nasal Cannula (HFNC): Non-invasive positive pressure ventilation
  High flow nasal cannula (HFNC): Non-invasive positive pressure ventilation Subjects: 27
- HFNC and External Nasal Dilator (END): high flow nasal cannula and external nasal dilator
  External nasal dilator (END): Applying External nasal dilator as adjuvant to high flow oxygen
  High flow nasal cannula (HFNC): Non-invasive positive pressure ventilation Subjects: 28
Period: Overall Study
Arm/Group | High Flow Nasal Cannula (HFNC) | HFNC and External Nasal Dilator (END)
Started | 27 | 28
Completed | 27 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Flow Nasal Cannula (HFNC) | HFNC and External Nasal Dilator (END) | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 28 | 55
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: months] | 10.31 [0 to 36] | 11.36 [0 to 36] | 10.8 [0 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 10 | 13 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 23 | 24 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change of Respiratory Status Using the Modified Bronchiolitis Severity Score, in Children Using External Nasal Dilators as an Adjuvant to High Flow Nasal Cannula Oxygen Therapy Compared to Those Receiving High Flow Nasal Cannula Therapy Alone
Description: Change of respiratory status using the Modified Bronchiolitis Severity Score in children using External Nasal Dilators as an adjuvant to High Flow Nasal Cannula oxygen therapy compared to those receiving High Flow Nasal Cannula therapy alone - shows that there is change in respiratory parameters, with positive number reflecting increases, and negative numbers reflecting decreases in number Modified Bronchiolitis Severity Score is measured by combining the individual score for five respiratory parameters (respiratory rate, breath sounds, work of breathing, oxygen saturation, mental status); score for each parameter ranges from 0-3; final score of each parameter is measured by adding them up; and so MBSS score ranges from 0-15; higher the score, worse the clinical status)
Time Frame: Change from baseline to time of hospital discharge, no greater than 1 month
Measure: Mean (Full Range); unit: number/score
Groups:
- High Flow Nasal Cannula (HFNC): Non-invasive positive pressure ventilation
  High flow nasal cannula (HFNC): Non-invasive positive pressure ventilation Higher MBSS
- HFNC and External Nasal Dilator (END): high flow nasal cannula and external nasal dilator
  External nasal dilator (END): Applying External nasal dilator as adjuvant to high flow oxygen
  High flow nasal cannula (HFNC): Non-invasive positive pressure ventilation Lower MBSS
Arm/Group | High Flow Nasal Cannula (HFNC) | HFNC and External Nasal Dilator (END)
Number analyzed (Participants) | 27 | 28
number/score | 1 [0 to 15] | 10 [0 to 15]

2. Secondary Outcome: Time Between Admission to Pediatric ICU to Discharge From Pediatric ICU
Description: Actual length of stay in pediatric ICU from admission to discharge
Time Frame: From subject enrollment to hospital discharge, not >170 hr
Measure: Median (Full Range); unit: hours
Groups:
- HFNC Group: High flow nasal cannula alone without external nasal dilator
- HFNC With END: High flow nasal cannula with external nasal dilator
Arm/Group | HFNC Group | HFNC With END
Number analyzed (Participants) | 27 | 28
hours | 73.5 [55.5 to 162] | 93.5 [54.5 to 135.5]

ADVERSE EVENTS:
Time Frame: Time period between between subject enrollment to hospital discharge not more than 1month
Description: None in both groups
Groups:
- High Flow Nasal Cannula (HFNC): Non-invasive positive pressure ventilation
  High flow nasal cannula (HFNC): Non-invasive positive pressure ventilation No adverse events
- HFNC and External Nasal Dilator (END): high flow nasal cannula and external nasal dilator
  External nasal dilator (END): Applying External nasal dilator as adjuvant to high flow oxygen
  High flow nasal cannula (HFNC): Non-invasive positive pressure ventilation No adverse events
Arm/Group | High Flow Nasal Cannula (HFNC) | HFNC and External Nasal Dilator (END)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 0/27 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No